CLINICAL TRIAL: NCT00859885
Title: Secondary Stroke Prevention In Patients With Patent Foramen Ovale: International PFO Consortium
Brief Title: International PFO Consortium
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University Hospital, Basel, Switzerland (Other); University of Lausanne Hospitals (Other); University Hospital, Geneva (Other); University Hospital, Zürich (Other); Triemli Hospital (Other); Cantonal Hospital of Aarau, Switzerland (Other); Alfried-Krupp Krankenhaus of Essen, Germany (Unknown); University Hospital, Essen (Other); Klinikum Worms (Other); Tufts Medical Center (Other); Baystate Medical Center (Other); East Medical Center Tyler, Texas (Unknown); Universitaire Ziekenhuizen KU Leuven (Other); Ammerland Klinik GmbH, Westerstede, Germany (Unknown); University Hospital, Ghent (Other); Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Prof. Dr. med. Krassen Nedeltchev, University of Bern and Triemli Hospital Zurich
Other Study IDs: 117/08
Record Dates: First submitted 2009-03-06; First posted 2009-03-11 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Stroke; Transient Ischemic Attack
Keywords: patent foramen ovale; ischemic stroke; transient ischemic attack; secondary prevention; medical treatment; percutaneous device closure
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient; Foramen Ovale, Patent; Ischemic Stroke | interventions — Aspirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients who receive antithrombotic treatment only
  Interventions: Drug: Antithrombotic treatment
- 2: Patients who undergo percutaneous device closure
  Interventions: Device: percutaneous device closure of PFO

INTERVENTIONS:
Drug: Antithrombotic treatment — antiplatelets, anticoagulants
  Other Names: aspirin
  Groups: 1
Device: percutaneous device closure of PFO — umbrella device for PFO closure
  Other Names: clopidogrel
  Groups: 2

SUMMARY:
The prevalence of patent foramen ovale (PFO) is about 25% in the general population and approximately 40% in patients who have ischemic stroke of unknown cause (cryptogenic stroke). Given the large number of asymptomatic patients, no primary prevention is currently recommended. On the contrary, secondary prevention is very important. Prospective studies have shown that antithrombotic treatment (ATT) with aspirin or warfarin appears to negate the risk of recurrent stroke associated with a PFO. Patients with spontaneous or large right-to-left shunts (RLS), those with a coinciding atrial septal aneurysm (ASA) or multiple ischemic events prior to the PFO diagnosis may still be at increased risk of stroke recurrence despite ATT. Percutaneous device closure (PDC) is a challenging alternative to ATT. Several studies reported 0% to 3.4% annual recurrence rates of stroke or TIA in patients treated by PDC. To date, there is no data from randomized controlled trials (RCT) comparing the risk of stroke recurrence after PDC with that under ATT only. The results from ongoing RCTs are not to be awaited in the near future, mainly due to low enrolment and event rates. Alternative data-gathering strategies such as multicenter registries are needed to overcome the low recruitment rates. The aim of the present study is to compare the risk of recurrent stroke and TIA in patients with PFO and otherwise unexplained stroke who undergo PDC or receive ATT.

DETAILED DESCRIPTION:
Background

The prevalence of patent foramen ovale (PFO) is about 25% in the general population and approximately 40% in patients who have ischemic stroke of unknown cause (cryptogenic stroke). Given the large number of asymptomatic patients, no primary prevention is currently recommended. On the contrary, secondary prevention is very important. Prospective studies have shown that antithrombotic treatment (ATT) with aspirin or warfarin appears to negate the risk of recurrent stroke associated with a PFO. Patients with spontaneous or large right-to-left shunts (RLS), those with a coinciding atrial septal aneurysm (ASA) or multiple ischemic events prior to the PFO diagnosis may still be at increased risk of stroke recurrence despite ATT. Percutaneous device closure (PDC) is a challenging alternative to ATT. Several studies reported 0% to 3.4% annual recurrence rates of stroke or TIA in patients treated by PDC. To date, there is no data from randomized controlled trials (RCT) comparing the risk of stroke recurrence after PDC with that under ATT only. The results from ongoing RCTs are not to be awaited in the near future, mainly due to low enrolment and event rates. Even if RCTs are completed successfully, statistical differences may remain undetected with the planned sample sizes. Alternative data-gathering strategies such as multicenter registries are needed to overcome the low recruitment rates.

Objective

1) To compare the risk of recurrent stroke and TIA in patients aged ≤ 55 years with PFO and otherwise unexplained stroke who undergo PDC or receive ATT only; 2) To assess the etiological role of PFO for stroke/TIA in patients aged > 55 years; 3) To assess the risk of recurrent stroke/TIA in "high-risk" PFO patients (i.e. those with spontaneous (at rest) or large RLS, coinciding ASA, or multiple previous cerebrovascular events).

Methods

Multicenter prospective non-randomized study with scheduled 3-years follow-up of patients with PFO and ischemic stroke or TIA. Participating centers: Swiss University Hospitals of Basel, Bern, Geneva, Lausanne and Zurich, the Cantonal Hospital of Aarau, the Triemli Hospital, the Alfried-Krupp Krankenhaus of Essen, the University Hospital of Essen, the Klinikum Worms gGmbH, Tufts Medical Center, Baystate Medical Center, the East Medical Center Tyler, and the University Hospital of Leuven.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Diagnosis of PFO established by transesophageal echocardiography (TEE)
* Ischemic stroke or transient ischemic attack within the previous 6 months

Exclusion Criteria

* Non-vascular origin of the neurological symptoms after brain imaging (CT scan or MRI)
* Comorbid condition that would interfere with the study
* Pregnancy
* History of intracranial bleeding, confirmed arterio-venous malformation, aneurysm or uncontrolled coagulopathy
* Contraindications for TEE, echocardiographic or iodine contrast media

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ischemic stroke or transient ischemic attacks, in whom a patent foramen ovale has been diagnosed by means of a transesophageal echocardiography
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2008-09-08 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
proportion of patients free of any stroke (including fatal stroke) or TIA | 3 years

SECONDARY OUTCOMES:
influence of gender, age, spontaneous or large shunt, coincidence of an atrial septum aneurysma | 3 years
influence of competitive causes of stroke | 3 years
frequency of residual shunt, (in)correct device position, need for implantation of second device and periprocedural complications | 30 days and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Krassen Nedeltchev, MD, Principal Investigator — Kantonsspital Aarau; Marie-Luise Mono, MD, Principal Investigator — Dep. of Neurology, Bern University Hospital, Bern; Marcel Arnold, MD, Study Director — University of Bern, Inselspital
Locations (18):
- United States (3):
  - Tufts Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - East Medical Center, Tyler, Texas
- Belgium (2):
  - University Hospital Gent, Ghent
  - Leuven University Hospital, Leuven
- Germany (4):
  - Alfried Krupp Hospital, Essen
  - Essen University Hospital, Essen
  - Ammerland Klinik GmbH, Westerstede
  - Klinikum Worms gGmbH, Worms
- Arcispedale Santa Maria Nuova, Department of Neurology, ASMN IRCCS, Reggio Emilia, Italy
- University Hospital Doctor Josep Trueta, Girona, Spain
- Switzerland (7):
  - Cantonal Hospital of Aarau, Aarau
  - Basel University Hospital, Basel
  - Department of Neurology, Bern University Hospital, Bern, Bern
  - Geneva University Hospital, Geneva
  - Lausanne University Hospital, Lausanne
  - Zürich Triemli Hospital, Zurich
  - Zürich University Hospital, Zurich